CLINICAL TRIAL: NCT01270178
Title: Prospective Trial of Entecavir for Chronic Hepatitis B in Hepatocellular Carcinoma Patients Underwent Radiofrequency Ablation Therapy
Brief Title: Entecavir for Chronic Hepatitis B in Hepatocellular Carcinoma Patients Underwent Radiofrequency Ablation Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Jaw-Ching Wu, M.D. Ph.D/ Attending Physician, Department of Medical Research and Education, Veterans General Hospital, Taipei, Taiwan
Other Study IDs: 20110103
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Hepatitis B; Hepatocellular Carcinoma
MeSH Terms: conditions — Hepatitis B, Chronic; Carcinoma, Hepatocellular | interventions — entecavir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Entecavir
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — film coated tablets / 0.5mg / once daily / 3 years

SUMMARY:
Persistent replication of HBV (47-55%) is frequently found in patients with HCC, which in turn leads to deterioration of liver reserve. Moreover, a large proportion of HCC patients who underwent curative therapy died from progressive liver decompensation rather than recurrence of cancer. It had been proved that anti-viral therapy for hepatitis C virus (HCV)-related HCC patients could reduce the rate of tumor recurrence after surgical resection.

This is a prospective study to evaluate the efficacy of ETV therapy in chronic hepatitis B patients after receiving RFA therapy for HCC.

ELIGIBILITY:
Inclusion Criteria:

* HCC diagnosed by pathology verification or in accordance with the guidelines of American Association for the Study of Liver Diseases published in 2010 (typical vascular pattern in computed tomography scan or magnetic resonance imaging study) ,
* Solitary tumor less than 5 cm in diameter or 2-3 tumors with the largest one no more than 3 cm in diameter,
* No extrahepatic metastasis,
* No radiological evidence of invasion into major portal vein or hepatic vein branches,
* Good liver reserve with Child-Pugh Class A or B,
* A platelet count of more than 50,000/mm3,
* Serum creatinine level ≤ 2 mg/dL,
* No previous treatment for HCC,
* Positive for serum hepatitis B surface antigen (HBsAg) for more than 6 months
* Positive serum HBV DNA using a Cobas Amplicor HBV monitor (Roche Diagnostic System, Basel, Switzerland).

Exclusion Criteria:

* Dual or multiple infections with hepatitis C virus, hepatitis D virus, or the human immunodeficiency virus,
* Other forms of liver disease such as alcoholic hepatitis, autoimmune hepatitis, Wilson's disease, hemochromatosis,
* Use of interferon alpha, thymosin or antiviral agents within 6 months preceding entry into the study,
* Women who are pregnant or nursing.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic hepatitis B patients received RFA therapy for HCC
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2011-01

PRIMARY OUTCOMES:
The survival rate and recurrence rate between patients receiving ETV therapy and those in historical control | 3 years

SECONDARY OUTCOMES:
HBV reactivation, incidence of ALT normalization, reduction of serum HBV DNA level, HBsAg loss and HBsAg seroconversion to anti-HBsAb, emergence of resistance. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan